CLINICAL TRIAL: NCT02846181
Title: A Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-SK-1405
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MO002A
Record Dates: First submitted 2016-07-11; First posted 2016-07-27 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-09

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

ARMS (1):
- Healthy (Experimental)
  Interventions: Drug: [14C]-SK-1405

INTERVENTIONS:
Drug: [14C]-SK-1405

SUMMARY:
The primary objectives of the study are:

* To assess the mass balance recovery after a single PO dose of [14C]-SK-1405
* To provide plasma, urine and faecal samples for metabolite profiling and structural identification

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 30 to 65 years of age
* Body mass index of 18.0 to 30.0 kg/m2
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Participation in a clinical research study within the 3 months prior to IMP dose
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* Subjects who have been dosed with SK-1405 in the past
* Subjects who are taking, or have taken, antiepileptic and/or antidepressant medication in the 6 months prior to dosing
* Subjects who are taking, or have taken, any prescribed medication in the 28 days prior to dosing, unless judged as not clinically significant by the investigator and sponsor
* Subjects who are taking, or have taken, any over-the-counter medication (with the exception of up to 2,000 mg/day paracetamol/acetaminophen) in the 7 days prior to dosing, unless judged as not clinically significant by the investigator and sponsor
* Use, during the 28 days prior to dosing, of any medicine or herbal remedy (such as St John's wort) known to induce or inhibit CYP enzymes, unless judged as not clinically significant by the investigator and sponsor
* History of any drug or alcohol abuse in the past 2 years
* History of clinically significant neurological conditions
* A QTcF >450 msec at screening, admission or pre-dose (as confirmed by a repeat ECG)
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months; this includes cigarettes, e-cigarettes and nicotine replacement products. A breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Subjects who have been enrolled in an ADME study in the last 12 months
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator, including AST, ALT or alkaline phosphatase >1.5 × upper limit of normal confirmed by repeat testing 18. Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation
* History of clinically significant psychiatric, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
* History of gastrointestinal surgery (except appendectomy) or any condition that may affect the absorption, distribution, metabolism or excretion of study drug in the opinion of the investigator
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy (including food or drug allergy) requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
* Donation or loss of greater than 400 mL of blood within the 3 months prior to IMP dose
* Subjects who have consumed St John's wort, red wine, Seville oranges, grapefruit or grapefruit juice within 7 days prior to dosing. Subjects must be willing to refrain from consuming such products until the last PK sample
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
14C radioactivity concentration excreted in urine | Every day for 14 days
14C radioactivity concentration excreted in faeces | Every day for 14 days
14C radioactivity concentration in whole blood | Every day for 14 days
14C radioactivity concentration in plasma | Every day for 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Ltd., Nottingham, United Kingdom